CLINICAL TRIAL: NCT00008489
Title: A Randomized Open-Label Trial Comparing the Tolerability of Videx EC Capsules to Videx Tablets in Adults With HIV Infection
Brief Title: Comparing Side Effects of Two Forms of Videx in HIV-Infected Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PharmaResearch (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 315A; BMS-006
Record Dates: First submitted 2001-08-30; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-01

CONDITIONS: HIV Infections
Keywords: Didanosine; Gastrointestinal System; Tablets; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Capsules
MeSH Terms: conditions — HIV Infections | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare gastrointestinal (stomach and intestines) side effects of 2 forms of Videx in HIV-infected patients.

Videx can be an effective anti-HIV treatment but many patients will not take the medication due to its side effects. Videx EC is a capsule form of the drug and may have fewer side effects. Also, patients would not have to take as many pills since patients taking Videx EC would have to take only 1 capsule per day instead of 2 tablets per day. This study will see if patients taking Videx EC have fewer side effects.

DETAILED DESCRIPTION:
Despite its therapeutic advantages and proven efficacy in the treatment of HIV-infected patients, didanosine may continue to be underutilized because many patients experience undesirable gastrointestinal (GI) side effects and palatability problems. Once-daily dosing with Videx EC is expected to improve patient adherence with possible improved palatability and remove the GI side effects associated with the buffers included in the tablet. Videx EC once-daily dosing would improve pill burden by decreasing from 2 tablets to 1 capsule per day. Therefore, Videx EC may represent a significant step toward achieving better patient satisfaction, improved regimen adherence, and optimal virologic outcomes with Videx-containing regimens.

Patients are randomized to either continue their current Videx tablet-containing regimen for an additional 2 weeks or replace their Videx tablets with Videx EC. Patients who remain on Videx tablets are switched to the EC formulation at Study Week 2 for the remaining 4 weeks of the study period. For patients who continue and successfully complete the Week 6 study visit, an optional extended dosing period is offered until Videx EC becomes commercially available or the study funder terminates the study. Blood specimens for safety evaluations and viral load are collected at Weeks 0, 1, 2, 4, and 6. For patients participating in the extended dosing period, the visit schedule is every 8 weeks. Symptom scores between the 2 treatment groups are compared, with the primary comparison occurring at the Week 2 visit. Analyses include changes in GSRS scores administered by clinician interview at each study visit. Assessment of GI symptoms, palatability features, dosing convenience, lifestyle effects, and Videx preference is evaluated by the patient. Adverse events are assessed objectively by the observations of both the investigator and the patient.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 16 years old (consent of parent or guardian required if under 18).
* Are taking a stable Videx-containing anti-HIV regimen, using Videx tablets either once or twice a day, for at least 2 weeks prior to the screening visit.
* Score 2 or higher on the GSRS questionnaire for 1 or more of the following symptoms at the first 2 study visits: abdominal pain, nausea and vomiting, borborygmus, abdominal distension, and loose stools.
* Agree to use an effective barrier method of birth control during the study.
* Are available for at least 8 weeks.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Are taking Videx in liquid form, nelfinavir, or amprenavir.
* Have a history of pancreatitis or gallstones.
* Abuse alcohol or require drugs which, in the opinion of the investigator, may increase the risk of pancreatitis.
* Have had treatment for an active opportunistic (AIDS-related) infection within 4 weeks of the screening visit. Patients with chronic candidiasis (yeast infection) or bacterial infection will be allowed.
* Are receiving or plan to receive chemotherapy for cancer.
* Plan to change their medications within 8 weeks following the screening visit.
* Are receiving investigational drugs or are participating in a clinical trial involving anti-HIV medications. Patients in Phase IV studies (studies that evaluate the long-term safety and effectiveness of a drug, usually after the drug has been approved by the FDA) may be eligible.
* Have an active, ongoing gastrointestinal disease or infection such as colitis, diverticulitis, Crohn's disease, peptic ulcer disease, giardiasis, or cryptosporidiosis.
* Are unable to take medications by mouth.
* Have severe diarrhea.
* Have peripheral neuropathy (a condition affecting the nervous system) or other condition or prior therapy that, in the opinion of the investigator, would affect the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Altamed Medical Health Services, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - Pacific Horizons Med Group, San Francisco, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Atlanta VA Med Ctr, Decatur, Georgia
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Park Nicollet Med Ctr / Hlth Education, Saint Louis Park, Minnesota
  - Treatment for Life Ctr, Brooklyn, New York
  - Jemsek Clinic, Huntersville, North Carolina
  - Bornemann Internal Medicine, Reading, Pennsylvania
  - Burnside Clinic, Columbia, South Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia